CLINICAL TRIAL: NCT06002477
Title: Attentional Mechanisms of Cognitive Compensation in Subjective Cognitive Decline
Brief Title: Attentional Mechanisms in SCD
Acronym: AMoCC-SCD
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Kimberly Albert, Research Assitant Professor, Psychiatry, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 230736
Record Dates: First submitted 2023-08-15; First posted 2023-08-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Subjective Cognitive Decline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anticholinergic Challenge (Experimental): All participants will receive oral mecamylamine for 1 day
  Interventions: Drug: Mecamylamine Challenge
- Placebo Challenge (Placebo Comparator): All participants will receive oral placebo for 1 day
  Interventions: Other: Placebo Comparator Challenge

INTERVENTIONS:
Drug: Mecamylamine Challenge — Mecamylamine 20 mg oral pill administered once
  Arms: Anticholinergic Challenge
Other: Placebo Comparator Challenge — Matching placebo oral pill administered once
  Arms: Placebo Challenge

SUMMARY:
This study will use an anticholinergic pharmacological probe to examine attention network function in SCD using EEG. The overall hypothesis is that in older adults with SCD, normal cognitive performance is maintained by compensatory attention network activity, supported by enhanced cholinergic function. The investigators anticipate that SCD will be associated with greater compensatory attention network activity and that disrupting this compensatory process through anticholinergic challenge will result in a greater negative effect on attentional performance (Attention Network Test, ANT) and attention network functioning (EEG) in older adults with greater subjective cognitive concern.

DETAILED DESCRIPTION:
Overview: Cognitively normal older adults with and without subjective cognitive decline (SCD) (n = 80) will complete two study visits that will be double blinded and randomized for anticholinergic challenge (mecamylamine or placebo). Drug challenge visits will include cognitive testing and an electroencephalography (EEG) session.

AIM 1: Test for anticholinergic effects on attentional network function by cognitive concern severity. Under anticholinergic challenge, compared to placebo, greater subjective cognitive concerns will be associated with…:

Hyp. 1a: greater reduction in orienting attention network activity (ERP amplitude for early attention orienting).

Hyp. 1b: greater negative change in orienting attention performance.

Screening Procedures:

We will assure participants do not have MCI using the MoCA and GDS. Participants scoring below 26 on the MoCA or above 3 on the GDS will be excluded.

Medical history and comorbidity will be quantified using the Cumulative Illness Rating Scale (CIRS) 90. Self-reported medical histories, and problem lists from electronic medical records will be reviewed for excluded medication and illness. Vital signs (weight, and height) will be assessed. Participants will complete an electrocardiogram and blood samples will be collected for a comprehensive metabolic panel and thyroid stimulating hormone levels.

All participants will be evaluated to exclude individuals with significant psychiatric symptoms using a partial Structured Clinical Interview for DSM-IV-TR (SCID). Participants will also complete the Beck Depression Rating Scale (BDI) and the Beck Anxiety Inventory (BAI). Participants scoring above a BDI of 7 or a BAI of 15 will be excluded.

Study Drug Administration: During challenge drug study visits, participants will receive double-blinded administration of study drug (20 mg oral mecamylamine) or placebo. The order of administration will be randomized across study days. Randomization and dispensing will be managed by VUMC Investigational Drug Services.

Mecamylamine is a centrally and peripherally active non-competitive antagonist of nicotine (and presumably acetylcholine) at C6 (ganglionic) type nicotinic receptors. Peak cognitive and physiologic effects occur by 2-3 hours and dissipate by 4-6 hours after oral administration. At the doses to be used in this study, the expected physiologic effects of mecamylamine include cycloplegia, mydriasis, drowsiness, partial amnesia, decreased bowel motility, tachycardia and decreased salivation. We have used mecamylamine extensively in clinical studies in identical doses to those proposed here.

EEG: Each participant will be tested individually in a quiet private room. EEG signals will be recorded using a 128-channel Geodesic sensor net (EGI, Inc., Eugene, OR). The net is made of Ag/AgCl-coated carbon electrodes embedded in soft electrolytic sponges and arranged into a net using elastomer strings. Each electrode is connected via carbon wiring to a high-impedance (1MOhm) low-noise amplifier that provides analogue-to-digital (A/D) conversion of the EEG signals.

Prior to application, the net is soaked in warm saline (KCl) solution. The electrode impedances will be kept at or below 40 kOhms. The use of high-impedance amplifiers minimizes any decrease in signal-to-noise ratio and allows collection of high-quality data without having to abrade the scalp, thus minimizing any discomfort and reducing infection risks. Tests of this system reported no significant signal loss over a range of EEG frequencies. Another advantage of this system is fast electrode application and impedance adjustments (< 10 minutes). The EEG signals will be sampled every 4ms with filters set at 0.1 Hz - 100 Hz. During data collection, all electrodes will be referred to vertex (Cz). EEG will be continuously monitored and during periods of motor activity or inattention, stimulus presentation will be suspended until behavior quiets. The entire recording session will last approximately 30 minutes.

Attention Network Test (15 minutes): A task designed to test three attentional networks: (1) alerting, (2) orienting, and (3) executive control. The ANT combines attentional and spatial cues with a flanker task (a central stimulus is flanked by distractors that can indicate the same or opposite response to the central stimulus). On each trial a spatial cue is presented, followed by an array of five arrows presented at either the top or the bottom of the computer screen. The participant must indicate the direction of the central arrow in the array of five.

The cue that precedes the arrows can be non-existent, a center cue, a double cue (one presented at each of the two possible target locations), or a spatial cue that deterministically indicates the upcoming target location. The alerting network contrasts performance (RT) with and without cues, the orienting network contrasts performance on the task with a spatial or neutral cue, and executive control (conflict) is measured by assessing interference from congruent and incongruent flankers.

Incidental Memory Task (8 minutes): A passive incidental visual memory paradigm will be used to evaluate changes in basic memory processes. Subjects will be asked to view a slide show of novel color photographs depicting complex natural scenes. A small subset of the stimuli will be presented repeatedly (x5) throughout the session; the rest will be shown once. To encourage attention to the stimulus sequence, 20 attention probes (yellow smiley face) will be presented throughout the test session and require a button press response.

Cognitive Assessments: Following the EEG session participants will complete cognitive assessments of memory, and psychomotor speed. Administration takes approximately 35 minutes. Our group has significant experience using these tests in older adult populations. Tests will be administered in the order indicated below. Participants will be trained to stable performance in the cognitive tasks to reduce learning effects on the repeated testing. Different versions of all tests will be used during training and at each administration to minimize the likelihood of carryover effects.

The tasks chosen are designed to assess a range of cognitive domains including multiple attention, and visual-spatial and verbal memory processes, as well as psychomotor speed. These tasks will be completed under placebo and anticholinergic challenge. The cognitive battery will assess 1)Attention Capacity: Multiple Object Tracking, Digit Symbol Coding; 2) Attention Vigilance: Critical Flicker Fusion; 3)Psychomotor Speed: Choice Reaction Time; 4)Visual Episodic Memory: Picture Sequence Memory Task (NIH Toolbox); 5)Verbal episodic Memory: Buschke Selective reminding Task; 6)Visual-Spatial Working Memory: Visual-Spatial N-Back. The time to complete the cognitive battery will be less than two hours which is well within the 4-6-hour duration of effect of 10 mg mecamylamine.

Statistical Analysis Plan:Power was calculated for the Aim1 primary outcome measure of correlation between CCI score and anticholinergic challenge effect on ANT orienting P1 amplitude. With a sample size of n = 80 and alpha = 0.05, for a weak moderate correlation (r = 0.40) we will have over 95% power. This sample size is also appropriate for the resting-state fMRI analyses.

AIM 1 examines anticholinergic challenge effects on:

Hyp 1a: Peak P1 amplitude in parietal regions for Orienting trials of the Attention Network Test (ANT)

The primary ANT ERP measure will be P1 amplitude for the orienting trials in parietal electrodes. The P1 ERP peak amplitude will be measured between 150 - 250 ms after spatial orienting cue onset. Peak P1 amplitude measured between 150 - 250 ms after the non-spatial cue will be used as the baseline P1 measure. Exploratory analyses will also examine peak P1 amplitude averaged across frontal electrodes and peak Executive P3 amplitude measured between 250 - 500 ms after executive incongruent target onset (compared to P3 amplitude for congruent targets).

Cognitive concern severity will be measured as the number of items endorsed on the 20 item Cognitive Change Index (CCI).

Hyp 1a will be analyzed using a linear mixed effects model analysis, with Orienting P1 amplitude as the dependent variable and drug challenge (mecamylamine or placebo), CCI score, and their interaction, as fixed factors.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 55
2. Montreal Cognitive Assessment (MoCA) > 25 AND Global Deterioration Scale (GDS) rating < 3
3. Non-smokers

Exclusion Criteria:

1. medical contraindications to the drug challenge
2. primary neurological disorder (such as stroke, epilepsy, etc.)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Peak P1 amplitude for Orienting | After administration of second drug challenge, approximately 72 hours
  Peak P1 amplitude in parietal regions for Orienting trials of the Attention Network Test (ANT) dyrung anticholinergic challenge

CONTACTS AND LOCATIONS:
Overall Officials: Paul Newhouse, MD, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No